CLINICAL TRIAL: NCT06395428
Title: Haloperidol for Pain Control in Patients With Acute Musculoskeletal Back Pain in the Emergency Department
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Western Michigan University School of Medicine (Other)
Collaborators: Bronson Methodist Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WMed-2024-1032
Record Dates: First submitted 2024-02-01; First posted 2024-05-02 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Back Pain; Chronic Pain
Keywords: Haloperidol; Chronic Pain; Back Pain
MeSH Terms: conditions — Back Pain; Chronic Pain | interventions — Haloperidol; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: This is a single-center prospective randomized double-blinded non-inferiority trial with potential assessment of superiority comparing haloperidol to ketorolac for the treatment of back pain.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment allocations will be revealed only after study completion, unless there is concern for a serious adverse event in which case treatment team and patient will be unblinded. Interim analysis will be performed at 34 participants to evaluate for effectiveness and power
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Haloperidol (Experimental): Haloperidol 5 mg IM haloperidol
  Interventions: Drug: Haloperidol
- Ketoralac (Active Comparator): Ketoralac 30 mg IM
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Haloperidol — Intramuscular injection of drug
  Other Names: Haldol
  Arms: Haloperidol
Drug: Ketorolac Tromethamine — Intramuscular injection of drug
  Other Names: Toradol
  Arms: Ketoralac

SUMMARY:
Single center, double-blind, randomized, controlled trial in patients who present to the emergency department (ED) with a chief complaint of back pain. A total of 150 patients age 18-65 presenting to the emergency department with chief complaint of backpain will be enrolled from April 2024 - April 2025. Patients will be randomized and symptom levels will be recorded at 30, 60, 90, minutes. Follow-up will be performed by telephone at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years old
* Presenting to the Bronson ED with a chief complaint of acute, non-traumatic back pain
* VAS score >5 cm

Exclusion Criteria:

* Back pain due to traumatic injury
* Experiencing saddle anesthesia
* Has bowel or bladder dysfunction
* Has an abnormal neurological exam
* Requires imaging in ED
* Has a Glascow coma score <15
* Has one or more abnormal vital signs:

HR>120, SBP>180 or <90, temperature >38°, O2 saturation<92%

* Has an allergy to ketorolac or haloperidol
* Has a known diagnosis of Lewy Body Dementia
* Has a known diagnosis of glaucoma.
* Is known to be pregnant or breastfeeding
* Is a prisoner or ward of the state
* Is unable to consent for themselves/ non-english speaking
* In the opinion of the attending physician or investigator the patient should not participate in the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 30, 60, and 90 minutes after drug administration
  Mean change in visual analog scale (VAS) of self-rated nausea severity

SECONDARY OUTCOMES:
Length of stay after enrollment | 24 hours
  Mean length of stay in minutes between the 2 groups will be assessed with a student's t test to assess for significant difference between groups
Need for rescue medications | 30, 60, and 90 minutes after drug administration
  Need for rescue medications will be a Boolean variable recorded in redcaps that will be qualitatively assessed to compare the number of patients in each group requiring rescue medication.
Patient Satisfaction | 24 hours after enrollment up to 1 week
  This will be assessed based on the follow-up question "would you receive this treatment again?" on the follow-up phone call. Number of patients in each group that answer yes to this question will be qualitatively discussed in the results.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica McCoy, MD, Principal Investigator — Western Michigan University Homer Stryker M.D. School of Medicine
Locations (1):
- Bronson Methodist Hospital, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The subject's info collected as part of the research, even if identifiers are removed, will not be used or distributed for future research studies.

REFERENCES:
- [Background] Silberstein SD, Peres MF, Hopkins MM, Shechter AL, Young WB, Rozen TD. Olanzapine in the treatment of refractory migraine and chronic daily headache. Headache. 2002 Jun;42(6):515-8. doi: 10.1046/j.1526-4610.2002.02126.x. PMID 12167140
- [Background] McCoy JJ, Aldy K, Arnall E, Petersen J. Treatment of Headache in the Emergency Department: Haloperidol in the Acute Setting (THE-HA Study): A Randomized Clinical Trial. J Emerg Med. 2020 Jul;59(1):12-20. doi: 10.1016/j.jemermed.2020.04.018. Epub 2020 May 10. PMID 32402480
- [Result] Todd KH, Ducharme J, Choiniere M, Crandall CS, Fosnocht DE, Homel P, Tanabe P; PEMI Study Group. Pain in the emergency department: results of the pain and emergency medicine initiative (PEMI) multicenter study. J Pain. 2007 Jun;8(6):460-6. doi: 10.1016/j.jpain.2006.12.005. Epub 2007 Feb 15. PMID 17306626
- [Result] Edwards J, Hayden J, Asbridge M, Gregoire B, Magee K. Prevalence of low back pain in emergency settings: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2017 Apr 4;18(1):143. doi: 10.1186/s12891-017-1511-7. PMID 28376873
- [Result] Kea B, Fu R, Lowe RA, Sun BC. Interpreting the National Hospital Ambulatory Medical Care Survey: United States Emergency Department Opioid Prescribing, 2006-2010. Acad Emerg Med. 2016 Feb;23(2):159-65. doi: 10.1111/acem.12862. Epub 2016 Jan 23. PMID 26802501
- [Result] Hoppe JA, Kim H, Heard K. Association of emergency department opioid initiation with recurrent opioid use. Ann Emerg Med. 2015 May;65(5):493-499.e4. doi: 10.1016/j.annemergmed.2014.11.015. Epub 2014 Dec 18. PMID 25534654
- [Result] Ruhm CJ. Geographic Variation in Opioid and Heroin Involved Drug Poisoning Mortality Rates. Am J Prev Med. 2017 Dec;53(6):745-753. doi: 10.1016/j.amepre.2017.06.009. Epub 2017 Aug 7. PMID 28797652
- [Result] Bertrand S, Meynet G, Taffe P, Della Santa V, Fishman D, Fournier Y, Frochaux V, Ribordy V, Rutschmann OT, Hugli O. Opiophobia in Emergency Department Healthcare Providers: A Survey in Western Switzerland. J Clin Med. 2021 Mar 25;10(7):1353. doi: 10.3390/jcm10071353. PMID 33805916
- [Result] Gueant S, Taleb A, Borel-Kuhner J, Cauterman M, Raphael M, Nathan G, Ricard-Hibon A. Quality of pain management in the emergency department: results of a multicentre prospective study. Eur J Anaesthesiol. 2011 Feb;28(2):97-105. doi: 10.1097/EJA.0b013e3283418fb0. PMID 21119516
- [Result] Duncan RW, Smith KL, Maguire M, Stader DE 3rd. Alternatives to opioids for pain management in the emergency department decreases opioid usage and maintains patient satisfaction. Am J Emerg Med. 2019 Jan;37(1):38-44. doi: 10.1016/j.ajem.2018.04.043. Epub 2018 Apr 22. PMID 29709398
- [Result] Rech MA, Griggs C, Lovett S, Motov S. Acute pain management in the Emergency Department: Use of multimodal and non-opioid analgesic treatment strategies. Am J Emerg Med. 2022 Aug;58:57-65. doi: 10.1016/j.ajem.2022.05.022. Epub 2022 May 22. PMID 35636044
- [Result] Verdu B, Decosterd I, Buclin T, Stiefel F, Berney A. Antidepressants for the treatment of chronic pain. Drugs. 2008;68(18):2611-32. doi: 10.2165/0003495-200868180-00007. PMID 19093703
- [Result] Kroeze WK, Hufeisen SJ, Popadak BA, Renock SM, Steinberg S, Ernsberger P, Jayathilake K, Meltzer HY, Roth BL. H1-histamine receptor affinity predicts short-term weight gain for typical and atypical antipsychotic drugs. Neuropsychopharmacology. 2003 Mar;28(3):519-26. doi: 10.1038/sj.npp.1300027. PMID 12629531
- [Result] Kiser RS, Cohen HM, Freedenfeld RN, Jewell C, Fuchs PN. Olanzapine for the treatment of fibromyalgia symptoms. J Pain Symptom Manage. 2001 Aug;22(2):704-8. doi: 10.1016/s0885-3924(01)00302-5. PMID 11495717
- [Result] Seidel S, Aigner M, Ossege M, Pernicka E, Wildner B, Sycha T. Antipsychotics for acute and chronic pain in adults. J Pain Symptom Manage. 2010 Apr;39(4):768-78. doi: 10.1016/j.jpainsymman.2009.09.008. Epub 2010 Mar 11. PMID 20226624
- [Result] Inayat F, Virk HU, Ullah W, Hussain Q. Is haloperidol the wonder drug for cannabinoid hyperemesis syndrome? BMJ Case Rep. 2017 Jan 4;2017:bcr2016218239. doi: 10.1136/bcr-2016-218239. PMID 28052951
- [Result] Cowling M, Covington S, Roehmer C, Musey P. Characterizing the role of haloperidol for analgesia in the Emergency Department. J Pain Manag. 2019;12(2):141-146. PMID 33193995
- See also: Haloperidol by Patriot Pharmaceuticals LLC / Johnson & Johnson Research & Development, LLC / Janssen Pharmaceutica NV / Janssen Pharmaceutica, NV HALOPERIDOL injection. — https://fda.report/DailyMed/c9d0d515-adb7-4f93-8363-0f11771321c9